CLINICAL TRIAL: NCT07255040
Title: A 24-Week, Randomised, Controlled, Examiner-blind, Clinical Study to Evaluate the Efficacy of an Experimental Stannous Fluoride Dentifrice in Improving Gingival Health and Reducing Plaque Accumulation
Brief Title: A Clinical Study to Evaluate the Effectiveness of an Experimental Toothpaste in Improving Gum Health and Reducing Plaque Accumulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400034
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Participants will be instructed to brush their teeth thoroughly with Test Dentifrice for at least one (timed) minute twice a day (morning and evening) for 24 weeks.
  Interventions: Drug: Test Dentifrice
- Reference Dentifrice (Positive Control) (Active Comparator): Participants will be instructed to brush their teeth thoroughly with Reference Dentifrice (Positive Control) for at least one (timed) minute twice a day (morning and evening) for 24 weeks.
  Interventions: Drug: Parodontax Complete Protection
- Reference Dentifrice (Negative Control) (Active Comparator): Participants will be instructed to brush their teeth thoroughly with Reference Dentifrice (Negative Control) for at least one (timed) minute twice a day (morning and evening) for 24 weeks.
  Interventions: Drug: Colgate Cavity Protection

INTERVENTIONS:
Drug: Test Dentifrice — Experimental dentifrice containing 0.454% w/w SnF2.
  Arms: Test Dentifrice
Drug: Parodontax Complete Protection — Marketed dentifrice containing 0.454% w/w SnF2.
  Arms: Reference Dentifrice (Positive Control)
Drug: Colgate Cavity Protection — Marketed regular fluoride dentifrice.
  Arms: Reference Dentifrice (Negative Control)

SUMMARY:
The aim of this 24-week clinical study is to evaluate the ability of an experimental dentifrice containing 0.454 percent (%) weight by weight (w/w) Stannous fluoride (SnF2); to improve gingival health, plaque reduction and prevention of plaque accumulation compared with a regular fluoride dentifrice (negative control) in participants with mild to moderate gingivitis.

DETAILED DESCRIPTION:
This will be a single-center, 24-week, randomized, controlled, single blind (examiner only), 3-treatment arms, parallel group, stratified study, to evaluate the efficacy of using an experimental dentifrice containing 0.454% w/w Stannous fluoride, twice daily in reducing gingivitis and plaque accumulation in a population with clinically measurable level of gingivitis. The clinical efficacy of the experimental dentifrice will be compared to a commercially available regular fluoride dentifrice as negative control. In addition, a marketed dentifrice containing 0.454% w/w SnF2 is included as positive control to provide a well-established benchmark. Approximately 300 participants (approximately 100 per group) will be randomized to ensure approximately 270 evaluable participants (approximately 90 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is at least 18 years old, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant 's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical, psychiatric condition or laboratory abnormality or any other clinical serious or unstable conditions (example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A female participant who is a pregnant (self-reported) or intending to become pregnant over the duration of the study or who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who is a current smoker or an ex-smoker (including vaping) who stopped within 6 months of Screening or who is using smokeless forms of tobacco (example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed with xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding (example, type 2 diabetes) or who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* Dental Exclusions:

  1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  2. A participant who has dentures (partial or full).
  3. A participant who has fixed orthodontic appliances or is undergoing active or recent (within 3 months of Screening) orthodontic treatment, which in the opinion of the investigator, could interfere with study procedures, assessments or outcomes.
  4. A participant who has other orthodontic devices (example, bands, fixed retainers, or removable retainers) that could, in the opinion of the investigator, interfere with study procedures, assessment or outcomes.
  5. A participant who has numerous restorations in a poor state of repair.
  6. A participant who has any dental condition (example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  7. A participant who has had dental prophylaxis within 12 weeks of Screening.
  8. A participant who has had teeth bleaching within 12 weeks of Screening.
  9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Bleeding Sites (Overall) at Week 24 | Week 24
  Number of bleeding sites will be assessed using the bleeding index (BI) assessment. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 millimeter (mm) into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. The number of bleeding sites for each participant will be calculated as the number of tooth sites with bleeding observed immediately on probing or within 30 seconds of probing.

SECONDARY OUTCOMES:
Number of Bleeding Sites (Overall) at Weeks 1, 4 and 12 | Weeks 1, 4 and 12
  Number of bleeding sites will be assessed using the BI assessment. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 mm into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. The number of bleeding sites for each participant will be calculated as the number of tooth sites with bleeding observed immediately on probing or within 30 seconds of probing.
Number of Bleeding Sites (Interproximal) at Weeks 1, 4 and 12 | Weeks 1, 4 and 12
  Number of bleeding sites will be assessed using the BI assessment. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 mm into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. The number of bleeding sites for each participant will be calculated as the number of tooth sites with bleeding observed immediately on probing or within 30 seconds of probing.
Number of Bleeding Sites (Interproximal) at Week 24 | Week 24
  Number of bleeding sites will be assessed using the BI assessment. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 mm into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. The number of bleeding sites for each participant will be calculated as the number of tooth sites with bleeding observed immediately on probing or within 30 seconds of probing.
Mean BI (Overall) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  The BI is an invasive assessment of gingival bleeding. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 mm into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. Gingival bleeding will be scored on a 3-points scale with scores ranging from 0 to 2, where 0=Absence of bleeding on probing, 1=Bleeding observed within 30 seconds of probing, 2=Bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Mean BI (Interproximal) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  The BI is an invasive assessment of gingival bleeding. BI will be assessed for all evaluable surfaces of the facial and lingual/palatal gingiva, six sites per tooth. The probe will be inserted approximately 1 mm into the gingival sulcus and moved around the tooth from the distal interproximal area to the mesial interproximal area, gently stretching the gingival epithelium. Gingival bleeding will be scored on a 3-points scale with scores ranging from 0 to 2, where 0=Absence of bleeding on probing, 1=Bleeding observed within 30 seconds of probing, 2=Bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Mean Modified Gingival Index (MGI) (Overall) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). The MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth. Three scores will be recorded buccally/labially and three scores lingually/palatally using a 5-point scale ranging from 0 to 4, where 0 = Absence of inflammation, 1= Mild inflammation: slight change in color, little change in texture of any portion of the marginal or papillary gingival unit, 2=Mild inflammation: criteria as [1] but involving the entire marginal or papillary gingival unit, 3=Moderate inflammation: glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, 4=Severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Mean MGI (Interproximal) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). The MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth. Three scores will be recorded buccally/labially and three scores lingually/palatally using a 5-point scale ranging from 0 to 4, where 0 = Absence of inflammation, 1= Mild inflammation: slight change in color, little change in texture of any portion of the marginal or papillary gingival unit, 2=Mild inflammation: criteria as [1] but involving the entire marginal or papillary gingival unit, 3=Moderate inflammation: glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, 4=Severe inflammation: marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Mean Turesky Plaque Index (TPI) (Overall) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  TPI will be used to assess plaque on all gradable teeth. The plaque will first be disclosed using a plaque disclosing dye solution. The TPI will be assessed on the facial and lingual surfaces of each scorable tooth. Three scores will be recorded buccally/labially and three scores lingually/palatally. Disclosed plaque will be scored on a scale ranging from 0-6, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering less than (<)1/3 of the tooth surface, 4=Plaque covering greater than or equal to (>=)1/3 but <2/3 of the tooth surface, 5=Plaque covering >=2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Mean TPI (Interproximal) at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  TPI will be used to assess plaque on all gradable teeth. The plaque will first be disclosed using a plaque disclosing dye solution. The TPI will be assessed on the facial and lingual surfaces of each scorable tooth. Three scores will be recorded buccally/labially and three scores lingually/palatally. Disclosed plaque will be scored on a scale ranging from 0-6, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4=Plaque covering >=1/3 but <2/3 of the tooth surface, 5=Plaque covering >=2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Change in Mean TPI From Pre to Post Single Brush at Baseline | Pre to Post Brushing at Baseline
  TPI will be used to assess plaque on all gradable teeth. The plaque will first be disclosed using a plaque disclosing dye solution. The TPI will be assessed on the facial and lingual surfaces of each scorable tooth. Three scores will be recorded buccally/labially and three scores lingually/palatally. Disclosed plaque will be scored on a scale ranging from 0-6, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3=Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4=Plaque covering >=1/3 but <2/3 of the tooth surface, 5=Plaque covering >=2/3 of the tooth surface. Lower score indicates improvement in the symptoms. Change in TPI will be calculated by subtracting pre brushing TPI score from post brushing TPI score at Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.